CLINICAL TRIAL: NCT04259437
Title: A Study to Evaluate the Gastrointestinal Tolerance and Acceptability of a High Energy, High Protein Low Volume Oral Nutritional Supplement in Adult Patients With or at Risk of Malnutrition
Brief Title: Gastrointestinal Tolerance of a Nutritional Supplement in Adult Patients With or at Risk of Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BL44
Record Dates: First submitted 2020-01-29; First posted 2020-02-06 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Gastro-Intestinal Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Protein, Energy Dense Nutritional Supplement (Experimental): 2 servings per day
  Interventions: Other: High Protein, Energy Dense Nutritional Supplement

INTERVENTIONS:
Other: High Protein, Energy Dense Nutritional Supplement — Ready to drink oral supplement

SUMMARY:
The purpose of this study is to evaluate the GI tolerance, palatability and compliance to a high protein energy-dense oral nutrition supplement in adult patients with or at risk of malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated informed consent form approved by Independent Ethics Committee and provided applicable privacy authorization prior to any participation in the study.
* Subject is considered malnourished or at risk for malnutrition
* Subject has normal GI function
* Subject requires oral nutritional supplementation ands is willing to comply with the study protocol

Exclusion Criteria:

* Subject has severe dementia, eating disorder, history of significant neurological or psychiatric disorder affecting abilities to answer questions, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Subject has a history of diabetes
* Subject is currently taking antibiotics or has taken antibiotics within 1 week prior to enrollment
* Subject has undergone major GI surgery less than 3 months prior to enrollment
* Subject has active malignant disease or was treated within the last 6 months for cancer
* Subject has immunodeficiency disorder
* Subject has had a myocardial infarction within the last 3 months prior to enrollment
* Subject is known to be allergic to intolerant to an ingredient found in the study product
* Subject has an aversion to the flavor of product being tested
* Subject has an obstruction of the GI tract precluding ingestion or absorption of the study product, inflammatory bowel disease, gastric esophageal reflux disease, short bowel syndrome, or other major gastro-intestinal disease-causing symptoms including but not limited to uncontrollable severe diarrhea, nausea, or vomiting
* Subject is taking medications/dietary supplements/substances that could profoundly modulate metabolism or affect gastrointestinal motility.
* Participation in another study that has not yet been approved as a concomitant study by the Sponsor.
* Subject has a clinical condition that is contraindicated with this product.
* Subject is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Tolerance | Day 1 to Day 7
  Subject completed Bristol Stool Type questionnaire; Stool is classified into 7 groups (Types 1-7) with Type 3-4 as ideal stools.
Nutritional Supplement Palatability | Day 1 to Day 7
  Subject completed 6, Likert Scale questions; 4 scaled in the negative direction; 2 scaled from Far Too to Not at all Enough
Nutritional Supplement Intake | Day 1 to Day 7
  Subject completed daily intake questionnaire including amount of Bottle 1 and Bottle 2 consumed
Nutritional Supplement Palatability | Day 7
  Subject completed 6, Likert Scale questions; 4 scaled in the negative direction; 2 scaled from Far Too to Not at all Enough for additional flavors

OTHER OUTCOMES:
Medications | Baseline to Day 7
  Subject reported medication usage
Weight | Baseline and Day 7
  For BMI Calculation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Camprubi Robles, PhD, Study Chair — Abbott
Locations (3):
- United Kingdom (3):
  - North Coast Medical Ltd, Newquay Health Centre, Newquay, Cornwall
  - Morrab Surgery, Penzance, Cornwall
  - The Adam Practice, Poole

IPD SHARING:
Plan to Share IPD: No